CLINICAL TRIAL: NCT03845712
Title: A Phase 2 Open-Label Study of Continuation Treatment With Combination Pyrimidine Nucleosides in Patients With Thymidine Kinase 2 Deficiency (TK2)
Brief Title: An Open-Label Study of Continuation Treatment With Combination Pyrimidine Nucleosides in Patients With TK2 Deficiency
Acronym: Continuation
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: UCB BIOSCIENCES, Inc. (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TK0102; 2018-004277-27 (EudraCT Number); U1111-1304-0423 (Other: World Health Organization (WHO)); 2023-510427-29 (Registry Identifier: EU Clinical Trials)
Record Dates: First submitted 2019-02-06; First posted 2019-02-19 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Thymidine Kinase 2 Deficiency
Keywords: Thymidine Kinase 2 Deficiency; TK2d; mitochondrial disorder; mitochondrial disease; Mitochondria; deoxycytidine and deoxythymidine; doxecitine and doxribtimine; MT1621; primary mitochondrial myopathy; mitochondrial depletion syndrome; Muscle weakness; Muscle atrophy; Loss of mobility
MeSH Terms: conditions — Mitochondrial Diseases; Muscle Weakness; Muscular Atrophy | interventions — Deoxycytidine; Thymidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- doxecitine and doxribtimine (Experimental): This is an open label study with all participants in a single arm. Study participants will take doxecitine and doxribtimine up to a maximum of 800 mg/kg/day (400 mg/kg/day doxecitine and 400 mg/kg/day doxiribtimine).
  Interventions: Drug: doxecitine and doxribtimine

INTERVENTIONS:
Drug: doxecitine and doxribtimine — Doxecitine and doxribtimine is administered orally in 3 equal doses given approximately 6 to 8 hours apart. Doxecitine and doxribtimine is administered with food.
  Other Names: MT1621; GMP grade dC/dT (deoxycytidine and deoxythymidine)

SUMMARY:
This is a Phase 2 prospective open-label treatment study of the safety and efficacy of doxecitine and doxribtimine in study participants with thymidine kinase 2 (TK2) deficiency who participated in the retrospective study MT-1621-101 [NCT03701568] or who were receiving nucleos(t)ide treatment and were approved by the Sponsor.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent by the parent(s) or legally authorized representative (LAR) and/or assent by the study participant (when applicable).
2. Confirmed genetic mutation in the TK2 gene.
3. Absence of other genetic disease or polygenic disease.
4. Current treatment with nucleos(t)ides for TK2 deficiency. Study participants who were not previously enrolled in MT-1621-101 [NCT03701568] will require Sponsor approval to ensure that collection of clinical and functional measurements prior to treatment are sufficient to serve as baseline assessments for purposes of evaluating safety and efficacy.
5. Female study participants must not be breastfeeding, have a negative pregnancy test at screening (females ≥10 years old), and have no intention to become pregnant during the course of the study. Female study participants who are of childbearing potential (ie, following menarche until ≥1 year post-menopausal if not anatomically and physiologically incapable of becoming pregnant) must agree and commit to the use of highly effective methods of birth control for the duration of the study and for 30 days after the end of the study. Acceptable methods are defined as those that result, alone or in combination, in a low failure rate (ie, <1% per year) when used consistently and correctly, such as surgical sterilization, an intrauterine device, or hormonal contraception in combination with a barrier method. In certain countries (if permitted by law), women of childbearing potential may instead agree to abide by heterosexual sexual abstinence during the study and for 30 days after the end of the study.
6. Male study participants with sexual partners should use condoms for the duration of the study and for 30 days after the last dose of study drug to prevent passing study drug to the partner in the ejaculate. Male participants should be advised not to donate sperm for 30 days after the last dose of study drug.
7. Willingness to maintain current treatment regimen and current exercise regimen for the duration of the clinical study.
8. Willingness to comply with the study protocol, including but not limited to, all study procedures, study visits, and study drug compliance.

Exclusion Criteria:

1. History of liver disease, or liver function test results (ALT, AST, or total bilirubin) ≥2× upper limit of normal without prior Sponsor approval.
2. Other significant medical condition that, in the opinion of the Investigator or Study Sponsor, may confound interpretation of the clinical course of TK2 deficiency.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2019-07-05 (Actual); Primary Completion 2026-02-19 (Estimated); Study Completion 2026-02-19 (Estimated)

PRIMARY OUTCOMES:
Safety as adverse events (AEs): number of participants who experience adverse events | Approximately 3 years
  Safety as determined by the number of participants who experience adverse events (AE), type of AE, severity of AE.
Safety as determined by laboratory measurements | Approximately 3 years
  Number of Participants Who Experience a Clinically Significant Change from Baseline in Clinical Laboratory Tests.
Safety as determined by electrocardiograms (ECGs) | Approximately 3 years
  Number of Participants Who Experience a Clinically Significant Change from Baseline ECG.

SECONDARY OUTCOMES:
Efficacy - Motor Function Assessments | Approximately 3 years
  Patient or physician reported achievement (capable) or loss (not capable) of gross motor milestones.
Efficacy - Respiratory Status | Approximately 3 years
  Pulmonary Function Tests (PFTs).
Efficacy - Growth/Nutrition | Approximately 3 years
  Growth in patients over time compared to normals using the WHO reference standards and expressed as Z scores.
Efficacy - Growth/Nutrition | Approximately 3 years
  Requirement for supplemental feeding/feeding tube within 1 patient over time and time to change of status of use of supplemental feeding/feeding tube (tube inserted for feeding use vs tube removed).
Maximum plasma concentration (Cmax) of deoxycytidine and deoxythymidine | Approximately 3 years
  PK of dC and dT (Cmax - peak plasma concentration)
Time to maximum plasma concentration (Tmax) of deoxycytidine and deoxythymidine | Approximately 3 years
  PK of dC and dT (Tmax - time to maximum plasma concentration)
AUC - area under the plasma concentration time curve of deoxycytidine and deoxythymidine | Approximately 3 years
  PK of dC and dT (AUC - area under the plasma concentration time curve)
Apparent elimination half-life (t1/2) of deoxycytidine and deoxythymidine | Approximately 3 years
  PK of dC and dT (t1/2 - apparent elimination half-life)
Biomarkers (plasma from blood) | Approximately 3 years
  Biomarkers which may be related to TK2 disease and/or drug treatment (eg, number of participants with normal vs abnormal creatine kinase measured in u/l compared to normal ranges).
Biomarkers (plasma from blood) | Approximately 3 years
  Biomarkers which may be related to TK2 disease and/or drug treatment (eg, number of participants with normal vs abnormal lactate levels measured in mmol/l compared to normal ranges).
Quality of life through patient questionnaire - Individualized Neuromuscular Quality of Life (INQoL) | Approximately 3 years
  INQOL Questionnaire with 15 questions in 3 sections about muscle weakness, pain, fatigue, locking of muscles, droopy eyelids, vision, swallowing, daily activity, independence, relationships, feelings, appearance, and treatment where patients aged 12 years and older rate how they feel and their muscles function to accomplish daily activities on a scale of 0 to 7, where lower values are generally associated with a better outcome.
Characterization of health care utilization | Approximately 3 years
Efficacy Assessment: Clinical Global Impression of Improvement (CGI-I) and Patient Global Impression of Improvement (PGI-I) | Approximately 3 years
  Clinical Global Impression of Improvement (CGI-I) completed by Investigator and Patient Global Impression of Improvement (PGI-I) completed by the patient/caregiver.

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273
Locations (8):
- Tk0102 1005, New York, New York, United States
- Israel (3):
  - Tk0102 4038, Haifa
  - Tk0102 4039, Holon
  - Tk0102 4037, Nehariya
- Spain (4):
  - Tk0102 3102, Barcelona
  - Tk0102 3121, Esplugues de Llobregat
  - Tk0102 3031, Madrid
  - Tk0102 3101, Seville

IPD SHARING:
Plan to Share IPD: Yes
Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe, or global development is discontinued, and 18 months after trial completion. Investigators may request access to anonymized individual patient-level data and redacted trial documents which may include: analysis-ready datasets, study protocol, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed. All documents are available in English only, for a prespecified time, typically 12 months, on a password protected portal. This plan may change if the risk of re-identifying trial participants is determined to be too high after the trial is completed; in this case and to protect participants, individual patient-level data would not be made available.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe or global development is discontinued, and 18 months after trial completion.
Access Criteria: Qualified researchers may request access to anonymized IPD and redacted study documents which may include: raw datasets, analysis-ready datasets, study protocol, blank case report form, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed. All documents are available in English only, for a pre-specified time, typically 12 months, on a password protected portal.
URL: https://www.Vivli.org

REFERENCES:
- [Derived] Hernandez-Voth A, Sayas Catalan J, Corral Blanco M, Castano Mendez A, Martin MA, De Fuenmayor Fernandez de la Hoz C, Villena Garrido V, Dominguez-Gonzalez C. Deoxynucleoside therapy for respiratory involvement in adult patients with thymidine kinase 2-deficient myopathy. BMJ Open Respir Res. 2020 Nov;7(1):e000774. doi: 10.1136/bmjresp-2020-000774. PMID 33246973